CLINICAL TRIAL: NCT06565156
Title: A Prospective, Multicenter, Randomized, Controlled Trial of Non-healing Diabetic Foot Ulcers Treated With Standard Care With or Without BR-AM
Brief Title: Non-healing Diabetic Foot Ulcers Treated With Standard Care With or Without BR-AM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioStem Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BR-AM-DFU-101
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-infected Diabetic Foot Ulcer; Diabetic Foot; Diabetic Wound; Diabetic Foot Ulcer; Non-ischemic Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To reduce bias in the determination of closure, an independent blinded reviewer will review the image obtained from the wound measurement device in each case where the Investigator determines the wound has achieved closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR-AM plus Standard Care (Experimental): All subjects in the treatment group will receive sponsor-approved standard of care. Standard of care is defined as:
  * Debridement,
  * Wound cleansing with a neutral, non-irritating and non-toxic solution,
  * Non-adherent wound contact layer, a foam pad, alginate or hydrofiber dressing for moderately draining wounds, a secondary retention bandage, and
  * An off-loading device. Using an appropriate size to cover the entire wound area, BR-AM should be applied directly to the wound surface following sharp debridement. It is recommended that the product be trimmed to fit the area of the wound with sterile scissors before application.
  Interventions: Other: BR-AM
- Standard Care (Active Comparator): All subjects in the control group will receive sponsor-approved standard of care. Standard of care is defined as:
  * Debridement,
  * Wound cleansing with a neutral, non-irritating and non-toxic solution,
  * Non-adherent wound contact layer, a foam pad, alginate or hydrofiber dressing for moderately draining wounds, a secondary retention bandage, and
  * An off-loading device.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: BR-AM — BR-AM is a single-layer amniotic membrane allograft. BR-AM is manufactured by BioStem Technologies, Inc. and is processed by the bioREtain method which, briefly, includes initial disinfection, processing with isotonic solutions, dehydration at 37-40°C and electron beam sterilization.
  Arms: BR-AM plus Standard Care
Other: Standard Care — Standard of care is defined as:
  * Debridement,
  * Wound cleansing with a neutral, non-irritating and non-toxic solution,
  * Non-adherent wound contact layer, a foam pad, alginate or hydrofiber dressing for moderately draining wounds, a secondary retention bandage, and
  * An off-loading device.
  Arms: Standard Care

SUMMARY:
This trial is a multicenter, randomized, controlled study designed to evaluate the safety and efficacy of BioREtain® Amniotic Membrane (BR-AM) plus standard of care versus standard of care only in the treatment of diabetic foot ulcers. The trial design will control potential variables that may affect the outcome between the treatment group and the control group by standardizing the requirements for debridement, wound dressings, and offloading. Weekly subject visits will help monitor compliance in wound care and off-loading, as well as to document when wound closure is achieved. The study will also implement the use of an electronic imaging and measurement device using a standardized protocol to ensure the measuring of the wound surface area and volume is accurate, highly reproducible, and minimally variable.

There will also be a crossover treatment phase for those patients that were relegated to standard care only. After their 12-week standard of care treatment phase and for only those subjects that did not achieve complete wound closure, will be allowed to crossover for an additional 12 weeks of treatment with the BR-AM product following the protocol and procedures set forth within this document.

DETAILED DESCRIPTION:
This study examines a patient population with a diabetic foot ulcer (DFU) having adequate perfusion without clinical signs and symptoms of infection. Historical data has demonstrated that around 30% of DFUs heal within 12 weeks using standard care alone. However, roughly half of patients suffering from DFUs require additional measures, including advanced therapy. It is hypothesized that weekly applications of the human placental allograft BR-AM applied to a nonhealing DFU will result in a higher rate of wounds showing complete healing within 12 weeks of initiating therapy, compared to standard care alone.

This study has a crossover period, where subjects on standard care alone who do not achieve complete healing within 12 weeks of initiating therapy will be allowed to crossover to receive BR-AC over 12 additional weeks, to evaluate if their wound can achieve complete healing.

A follow-up phase will commence for all subjects that achieve complete wound closure, which is designed to measure longevity and durability of the closed wound. This follow up period will consist of a four-week follow up with two visits at each two-week interval.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the informed consent form.
* Male or female patient at least 18 years of age or older, as of the date of the screening visit.
* Confirmed diagnosis of Type 1 or Type 2 Diabetes.
* Has a DFU that is located below the malleoli at least 1.0 cm2 or up to 20.0 cm2 when measured by the investigator staff at the screening visit using the eKare device post debridement.

  a. If more than one ulcer is present the selected target ulcer must be at least 2 cm from the nearest edge of any adjacent ulcers.
* The depth of the target foot ulcer is graded as Wagner Grade I or II, i.e., with no evidence of exposed muscle, tendon, bone, or joint capsule.
* The target ulcer is "chronic, hard-to-heal," defined as having a duration of > 4 weeks but ≤ 52 weeks at the time of the screening visit.
* Arterial supply adequacy to the foot with the target ulcer confirmed by any one of the following:

  1. Great toe pressure ≥ 40 mm/Hg
  2. Systolic blood pressure Ankle Brachial Index (ABI) in the range ≥ 0.70 ≤ 1.20
  3. TcPO2 ≥ 30 mmHg from the foot
  4. Toe Brachial Index or TBI ≥ 0.50
* Willing to follow all instructions given by the Investigator, return for all visits, and adhere to off-loading protocols while on the study.

Exclusion Criteria:

* Hemoglobin A1c (HbA1c) level is > 12% (108 mmol/mol).
* Chronic oral steroid use of > 7.5 mg daily within the previous 30 days preceding screening.
* Chronic oral or parenteral corticosteroids, or any cytotoxic agents within the previous 30 days preceding screening.
* Has tested positive for Human Immunodeficiency Virus (HIV) or has Acquired Immune Deficiency Syndrome (AIDS).
* Has malignancy or history of cancer in 5 years preceding the screening visit other than non-melanoma skin cancer.
* Pregnant women.
* Women of child-bearing potential who are unwilling to avoid pregnancy or use an effective form of birth control.
* Currently on dialysis or planning to start dialysis.
* Is currently enrolled or participated in another device, drug, or biological trial within 30 days of screening.
* Has used wound treatments with enzymes, growth factors, living skin, dermal substitutes including other amniotic or umbilical cord tissue therapies, or other advanced biological therapies within the last 30 days.
* Current use of topical anti-microbial or silver-containing products.
* Target ulcer is over an active or inactive Charcot deformity.
* The depth of the target ulcer is graded as Wagner Grade III or higher, i.e., with evidence of exposed muscle, tendon, bone, and/or joint capsule.
* Gangrene is present on any part of the affected foot.
* Current suspicion of osteomyelitis, cellulitis, or other clinical signs or symptoms of target ulcer infection.
* Any previous use of Vendaje®, Vendaje AC®, AmnioWrap2® applied to the target ulcer.

The following additional exclusion criteria should be reviewed for all subjects at the end of the screening run-in period prior to randomization for eligibility determination:

* The target ulcer has decreased > 30% in wound area post debridement at baseline following the two-week run-in period.
* Use of excluded concomitant medications, therapies, or procedures during the two-week run-in period.
* Has clinical signs or symptoms of infection within the target ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To determine whether DFUs treated with standard care plus BR-AM results in a higher probability of achieving complete wound closure compared to standard care alone. | over the 12-week treatment period
  Percentage of subjects with complete wound closure over the 12-week treatment period, defined as 100% reepithelialization

SECONDARY OUTCOMES:
To compare differences between treatment groups in proportions of wounds with complete wound closure, based on time in days to closure. | at 12 weeks
  Percent change from baseline in wound surface area (cm2) at 12-weeks post-randomization.
To compare differences between treatment groups in percent change in wound area (cm2). | at 12 weeks
  Percent change from baseline in wound surface area (cm2) at 12-weeks post-randomization.
To compare differences between treatment groups in percent change in wound volume (cm3). | at 12 weeks
  Percent change from baseline in wound volume (cm3) at 12-weeks post-randomization.
To determine the total number of applications of BR-AM needed to achieve complete wound closure. | over 12-weeks post-randomization
  Total number of applications of BR-AM to achieve complete wound closure over 12-weeks post-randomization.
To determine whether subjects that crossover and receive standard care plus BR-AM results in a higher probability of achieving complete wound closure over the 12 additional weeks versus standard care alone based on time in days to closure. | over an additional 12 weeks
  Time in days from Visit 18 to initial observation of wound closure (defined as 100% reepithelialization of the wound without drainage) over an additional 12 weeks (Visits 19-30), where healing has been confirmed at two visits two weeks apart.

OTHER OUTCOMES:
Number of participants that acquire clinical signs and symptoms of infections post-randomization | over 12-weeks post-randomization
  Differences in clinical signs and symptoms of infection from Visit 2 through end of study between the treatment groups
Proportion of subjects experiencing adverse events, by treatment group | over the 17-week study period
  Spontaneously reported and elicited adverse events, coded in MedDRA

CONTACTS AND LOCATIONS:
Overall Officials: Bert Slade, MD, Study Director — Independent
Locations (17):
- United States (17):
  - Site 17, Guntersville, Alabama
  - Site 22, Mesa, Arizona
  - Site 25, Tucson, Arizona
  - Site 19, Palmdale, California
  - Site 02, San Francisco, California
  - Site 01, Vista, California
  - Site 27, Coral Gables, Florida
  - Site 20, Deerfield Beach, Florida
  - Site 28, DeLand, Florida
  - Site 23, Springfield, Illinois
  - Site 18, Boston, Massachusetts
  - Site 26, Detroit, Michigan
  - Site 16, Lake Success, New York
  - Site 15, Chapel Hill, North Carolina
  - Site 29, Brownsville, Texas
  - Site 21, Burleson, Texas
  - Site 24, San Antonio, Texas